CLINICAL TRIAL: NCT06031714
Title: "Study of CCR Receptor Overexpression in Fetal Microchimeric Cells: Proof of Concept Before a Potential Clinical Trial"
Brief Title: Fetal Cell Receptors Repertoire
Acronym: MoreCCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230731; 2023-A00404-41 (Other: ANSM)
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Venous Ulcer; Sickle Cell Ulcer; Diabetic Ulcer; Post-partum Women; Mixed Ulcer
Keywords: Microchimerism; Foetal stem cells; Receptors
MeSH Terms: conditions — Varicose Ulcer | interventions — Blood Specimen Collection; Interviews as Topic; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients (Other): Patients who have had at least one pregnancy and have a venous ulcer, diabetic ulcer or sickle cell ulcer
  Interventions: Other: Saliva sampling; Other: Blood sampling; Other: Interviews; Other: Clinical examination
- Patient "Controls group " (Other): Post-partum women of the same age but without wounds.
  Interventions: Other: Saliva sampling; Other: Blood sampling; Other: Interviews; Other: Clinical examination
- Children (Other)
  Interventions: Other: Saliva sampling

INTERVENTIONS:
Other: Saliva sampling — HLA genotyping. The technique should allow to identify, for children's, a paternal HLA antigen not shared with the mothers.
Other: Blood sampling — Maternal Blood samples will be incubated with the appropriate antibody, targeting the microchimeric fetal cells of each patient, as well as with a cell viability marker (DAPI). The samples were then be processed through the BD FACS Aria III to sort the fetal cells,
  The following steps - RNA extraction, quality control, retrotranscription, preparation of the library, sequencing and transcriptomic analysis - will be carried out according to the Smart-seq3 protocol. The data will be sent for in-depth analysis and confirmation of the results. Additional functional experiments may also be carried out.
  Arms: Patient "Controls group "; Patients
Other: Interviews — V2 and/or V3
  Arms: Patient "Controls group "; Patients
Other: Clinical examination — V2 and/or V3
  Arms: Patient "Controls group "; Patients

SUMMARY:
The purpose of this study is to describe the transcriptomic profile of foetal cells in post-partum and more specifically to determine which chemokine receptors are overexpressed in foetal cells in post-partum women with wounds To do so, the investigators will isolate foetal cells from the peripheral blood of healthy controls post partum women as well as from post partum women with skin ulcers and then perform RNA sequencing.

DETAILED DESCRIPTION:
The aim of regenerative medicine is to repair damaged tissue using different sources of autologous or heterologous stem cells. These cells are then cultured to achieve amplification and differentiation adapted to the cell type of the organ to be repaired. These methods are potentially effective, but involve risks and limitations, in particular the risks of genetic modifications during culture or contamination by residual ES or iPS cells. Immunosuppressive treatment is also necessary if the source of stem cells is allogeneic. Finally, implantation of this type of culture may also be unsuccessful.

Our team is seeking for an alternative strategy to these methods. This relies on the presence of a niche of foetal cells transferred during pregnancy that persist after delivery. In fact, all mammalian pregnancies lead to foetal-maternal cell transfer. The foetal cells -transferred to the maternal circulation- contain different types of stem cells that will remain in the maternal bone marrow and persist there for the rest of the mother's life. The team has shown that in the event of cutaneous wounds in post-gestational mice, a population of CD11b+ CD34+ CD31+ foetal progenitors was recruited from the maternal bone marrow to the cutaneous granulation tissue. These cells over-express the chemokine receptor CCR2 compared with their adult counterparts. Consequently, the injection of low, so-called physiological, doses of the CCL2 chemokine subcutaneously into wounds accelerates normal wound healing and restores delayed healing in two pathological models. This pro-healing activity is linked to the specific recruitment of foetal stem cells to the site of injected wounds. These low doses of CCL2 never affected wound healing in virgin mice, confirming that this type of treatment does not alter the homeostasis of adult cells.

The therapeutic strategy the investigators are proposing, entitled "natural stem therapy", is based on this reservoir of foetal stem cells present in every woman who has had at least one pregnancy, i.e. more than 60% of adult women in western countries. In order to test the validity of this concept, it is important to ascertain the pathways by which foetal cells are chemoattracted in the human species, in particular the CCR2/CCL2 pathway.

ELIGIBILITY:
Inclusion Criteria:

Common criteria :

* Adult women,
* Post-partum: having been pregnant for any length of time,
* Having signed a free and informed consent form,
* Primiparous or multiparous,
* Affiliated to a health insurance

Patients :

- Patients with a venous, diabetic or sickle cell ulcer, or mixed ulcer

Control group patients :

* Volunteers,
* Age-matched,
* Without skin ulcers.

There are no specific criteria for children.

Exclusion Criteria:

* Minors (for patients)
* Under court protection, curatorship, guardianship (for patients)
* Immunocompromised patients for any reason whatsoever
* Refusal of consent
* Refusal of blood and/or saliva samples for themselves or a member of their family

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic analysis by single cell sequencing | Month 1 up to month 5
  Transcriptomic analysis by single cell RNA sequencing (Smart-seq3 protocol) of fetal cells sorted from peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Sélim ARACTINGI, MD, PHD, Study Director — Dermatology unit, Cochin Hospital - APHP
Locations (1):
- Dermatology unit - Cochin Hospital - APHP, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided